CLINICAL TRIAL: NCT00258609
Title: A 12-week Prospective, Double-blinded, Randomized, Multicenter Study of Low Dose and Medium Dose Botulinum Toxin Type A (Dysport® ) Injection for Migraine Prophylaxis.
Brief Title: Dysport® In Migraine Without Aura Prophylaxis : DIMWAP Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Collaborators: Ipsen (Industry); Chiang Mai University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: A-38-52120-007
Record Dates: First submitted 2005-11-23; First posted 2005-11-24 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Migraine Without Aura Prophylaxis
Keywords: Botulinum toxin type A,; Dysport®,Dysport; Migraine without aura,; Migraine prophylaxis.
MeSH Terms: conditions — Migraine without Aura | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

INTERVENTIONS:
Drug: Botulinum Toxin type A (Dysport ® ) IM/SC 6-sites pericranial injection

SUMMARY:
The purpose of this study is to determine whether 120 Unit, and 240 unit of botulinum toxin A are effective in the treatment of migraine without aura prophylaxis.

DETAILED DESCRIPTION:
This is a 12-week, prospective double-blinded, randomized, multicenter study of placebo, 120 Unit, and 240 unit of botulinum toxin A ( Dysport ® ) injection for patient with a diagnosis of Migraine without aura according to International Headache Society criteria. It is designed to evaluate the efficacy, safety, tolerability and optimum dose of Botulinum toxin type A (Dysport ®)injection for migraine without aura prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

• The patient must give written (personally signed and dated) informed consent before completing any study-related procedure, which means any assessment or evaluation that would not have formed part of the normal medical care of the patient.• Able to give written inform consent and have a copied one.• Male or female patient age 18 - 65.• Patients are fulfil the International Headache Society diagnostic criteria for migraine• Patients experience an average of 2 to 8 migraine attacks per month over the 3 months and if they recorded 2 to 8 migraine attacks during the screening period. • Patients with prophylactic treatment for migraine have been unchanged for 3 months. • Able to continuation anti - migraine drugs.• Female patient in good general health who is potentially fertile and sexually active must be instructed by the investigator to avoid pregnancy during the study by condom or other contraceptive measure and has negative urine pregnancy test. (if possible at each visit a control of the urine pregnancy test will be performed).• Patients have to judge reliable for medication compliance and recording the effects of medication, as well as clearly motivated to obtain benefit from treatment. • The normal physical and neurological examinations during the whole study period. • Normal result for haematology test • Liver transaminase inferior than 2 upper normal values of the laboratory.

Exclusion Criteria:

• Patients are fulfil the international Headache Society criteria diagnostic for pure migraine with aura.• The patient is pregnant or lactating.• The patient is a female at risk of pregnancy during the study, not taking adequate precautions against pregnancy.• The patient has a known hypersensitivity to any of the test materials or related compounds.• The patient is unable or unwilling to comply fully with the protocol.• The patient has received any unlicensed drug within the previous 6 months.• Treatment with investigational drug (s) within 6 months before the screening visit.• The patient has previously entered this study.• Patient with past history of predominant tension type headache, botulism, other neuromuscular disorder (e.g. myasthenia gravis, Lambert - Elton Syndrome)• Patient with significant medical / neurological / psychiatric disorders such as blood dyscrasia,thrombocytopenia, rheumatoid arthritis, congestive heart failure, coronary artery heart diseases, dementia, psychosis, major depression or other conditions which could influence the clinical trial. • History of drugs abuse (narcotic (s), cafergot, or others) or drug (botulinum toxin type A) allergy.• Treatment with BTX A within 6 month Treatment or any medical condition that may have put the participant at risk with exposure to BTX-A (neuromuscular disorders, aminoglycoside antibiotics, curare-like agents).• History of migrainous infarction, hemiplegic migraine.• Unable to fill patient diary at home during migraine attack.• Patient who plan to schedule elective surgery during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128
Dates: Start 2003-02; Study Completion 2004-06

PRIMARY OUTCOMES:
Mean change from baseline of Area undercurve of headache diary ( total headache score).
Mean change from baseline of total duration of migraine attack( hours) in 4 weeks.
Mean change from baseline of migraine frequency

SECONDARY OUTCOMES:
MIDAS score, SF36

CONTACTS AND LOCATIONS:
Overall Officials: Siwaporn Chankrachang, MD, Principal Investigator — Northern Neurological Center, Faculty of Medicine,Chiang Mai University
Locations (6):
- Thailand (6):
  - Division of Neurology, Department of Medicine, Bhumipol Hospital., Bangkok
  - Division of Neurology, Department of Medicine, Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok
  - Division of Neurology, Department of Medicine, Pramongkutklao Hospital, Bangkok
  - Division of Neurology, Prasart Neurological Institute, Public Health Ministry., Bangkok
  - Northern Neurological Center, Faculty of Medicine, Chiang Mai University, Chiang Mai
  - Department of Medicine, Sappasithiprasong Hospital, Public Health Ministry, Ubonratchatani

REFERENCES:
- [Background] Silberstein S, Mathew N, Saper J, Jenkins S. Botulinum toxin type A as a migraine preventive treatment. For the BOTOX Migraine Clinical Research Group. Headache. 2000 Jun;40(6):445-50. doi: 10.1046/j.1526-4610.2000.00066.x. PMID 10849039
- [Background] Evers S, Vollmer-Haase J, Schwaag S, Rahmann A, Husstedt IW, Frese A. Botulinum toxin A in the prophylactic treatment of migraine--a randomized, double-blind, placebo-controlled study. Cephalalgia. 2004 Oct;24(10):838-43. doi: 10.1111/j.1468-2982.2004.00754.x. PMID 15377314
- [Background] Tepper SJ, Bigal ME, Sheftell FD, Rapoport AM. Botulinum neurotoxin type A in the preventive treatment of refractory headache: a review of 100 consecutive cases. Headache. 2004 Sep;44(8):794-800. doi: 10.1111/j.1526-4610.2004.04147.x. PMID 15330826
- [Background] Turton K, Chaddock JA, Acharya KR. Botulinum and tetanus neurotoxins: structure, function and therapeutic utility. Trends Biochem Sci. 2002 Nov;27(11):552-8. doi: 10.1016/s0968-0004(02)02177-1. PMID 12417130
- [Background] Brin MF. Botulinum toxin: chemistry, pharmacology, toxicity, and immunology. Muscle Nerve Suppl. 1997;6:S146-68. PMID 9826987
- [Background] Cui M, Khanijou S, Rubino J, Aoki KR. Subcutaneous administration of botulinum toxin A reduces formalin-induced pain. Pain. 2004 Jan;107(1-2):125-33. doi: 10.1016/j.pain.2003.10.008. PMID 14715398
- [Background] Borodic GE, Acquadro M, Johnson EA. Botulinum toxin therapy for pain and inflammatory disorders: mechanisms and therapeutic effects. Expert Opin Investig Drugs. 2001 Aug;10(8):1531-44. doi: 10.1517/13543784.10.8.1531. PMID 11772268
- [Background] Arezzo JC. Possible mechanisms for the effects of botulinum toxin on pain. Clin J Pain. 2002 Nov-Dec;18(6 Suppl):S125-32. doi: 10.1097/00002508-200211001-00003. PMID 12569959
- [Background] Kramer HH, Angerer C, Erbguth F, Schmelz M, Birklein F. Botulinum Toxin A reduces neurogenic flare but has almost no effect on pain and hyperalgesia in human skin. J Neurol. 2003 Feb;250(2):188-93. doi: 10.1007/s00415-003-0971-x. PMID 12574949
- [Background] Blersch W, Schulte-Mattler WJ, Przywara S, May A, Bigalke H, Wohlfarth K. Botulinum toxin A and the cutaneous nociception in humans: a prospective, double-blind, placebo-controlled, randomized study. J Neurol Sci. 2002 Dec 15;205(1):59-63. doi: 10.1016/s0022-510x(02)00313-1. PMID 12409185
- [Background] Caputi CA. Effectiveness of BoNT-A in the treatment of migraine and its ability to repress CGRP release. Headache. 2004 Sep;44(8):837-8. doi: 10.1111/j.1526-4610.2004.04158_1.x. No abstract available. PMID 15330838
- [Background] Smuts JA, Schultz D, Barnard A. Mechanism of action of botulinum toxin type A in migraine prevention: a pilot study. Headache. 2004 Sep;44(8):801-5. doi: 10.1111/j.1526-4610.2004.04148.x. PMID 15330827
- [Background] Durham PL, Cady R, Cady R. Regulation of calcitonin gene-related peptide secretion from trigeminal nerve cells by botulinum toxin type A: implications for migraine therapy. Headache. 2004 Jan;44(1):35-42; discussion 42-3. doi: 10.1111/j.1526-4610.2004.04007.x. PMID 14979881
- [Background] Silberstein SD. Review of botulinum toxin type A and its clinical applications in migraine headache. Expert Opin Pharmacother. 2001 Oct;2(10):1649-54. doi: 10.1517/14656566.2.10.1649. PMID 11825307
- [Background] Aoki KR. Evidence for antinociceptive activity of botulinum toxin type A in pain management. Headache. 2003 Jul-Aug;43 Suppl 1:S9-15. doi: 10.1046/j.1526-4610.43.7s.3.x. PMID 12887389
- [Background] Blumenfeld AM, Dodick DW, Silberstein SD. Botulinum neurotoxin for the treatment of migraine and other primary headache disorders. Dermatol Clin. 2004 Apr;22(2):167-75. doi: 10.1016/s0733-8635(03)00105-0. PMID 15222577
- [Background] Gobel H. Botulinum toxin in migraine prophylaxis. J Neurol. 2004 Feb;251 Suppl 1:I8-11. doi: 10.1007/s00415-004-1103-y. PMID 14991336
- [Background] Evers S, Rahmann A, Vollmer-Haase J, Husstedt IW. Treatment of headache with botulinum toxin A--a review according to evidence-based medicine criteria. Cephalalgia. 2002 Nov;22(9):699-710. doi: 10.1046/j.1468-2982.2002.00390.x. PMID 12421155
- [Background] Chankrachang S, Arayawichanont A, Poungvarin N, Nidhinandana S, Boonkongchuen P, Towanabut S, Sithinamsuwan P, Kongsaengdao S. Prophylactic botulinum type A toxin complex (Dysport(R)) for migraine without aura. Headache. 2011 Jan;51(1):52-63. doi: 10.1111/j.1526-4610.2010.01807.x. Epub 2010 Nov 16. PMID 21083558